CLINICAL TRIAL: NCT00367146
Title: MMF After Pediatric Liver Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hannover Medical School (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHH3474MMF
Record Dates: First submitted 2006-08-21; First posted 2006-08-22 (Estimated); Last update posted 2011-05-20 (Estimated); Status verified 2007-07

CONDITIONS: Liver Transplantation; Chronic Kidney Disease
Keywords: liver transplantation; children; immunosuppression; mycophenolatmofetil; calcineurin inhibitor; kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: MMF

SUMMARY:
The use of CNIs (CSA or FK) as primary immunosuppressive drugs after pediatric liver transplantation is one of the main causes of chronic kidney disease in these patients in the long term.

The study objective is the evaluation of safety of a modification in immunosuppression from a dual-immunosuppression (CSA or FK plus steroids) to a triple immunosuppression (MMF plus CSA (reduced dosage) plus steroids.

ELIGIBILITY:
Inclusion Criteria:

* patients after pediatric liver transplantation
* no acute rejections for the last half year

Exclusion Criteria:

* concomitant malign disease (e.g. ptld)
* neutropenia (granulocytes <1000/µl)
* systemic infection
* thrombopenia (<80/nl)

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2004-11; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
safety of a triple immunosuppression (MMF/CSA/Steroids)regarding the number of acute rejections | 1, 3, 6, 9, 12, 24 month

SECONDARY OUTCOMES:
incidence of chronic kidney disease | 12, 24 month
incidence of infections | 1, 3, 6, 9, 12, 24 month
incidence of ptld (post transplant lymphoproliferative disease) | 1, 3, 6, 9, 12, 24 month

CONTACTS AND LOCATIONS:
Overall Officials: Michael Melter, PhD, MD, Principal Investigator — Hannover Medical School
Locations (1):
- Hannover medical School, Hanover, Germany